CLINICAL TRIAL: NCT03972930
Title: Phase 2 Trial of Hypofractionated Radiotherapy for Soft Tissue Sarcomas
Brief Title: Hypofractionated Radiotherapy for Soft Tissue Sarcomas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW18149; 2019-0360 (Other: Institutional Review Board); A533300 (Other: UW Madison); SMPH/HUMAN ONCOLOGY/HUMAN ONCO (Other: UW Madison); NCI-2019-03768 (Registry Identifier: NCI Trial ID); Protocol Version 5/5/2021 (Other: UW Madison)
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Soft Tissue Sarcoma
Keywords: Hypofractionated Radiotherapy
MeSH Terms: conditions — Sarcoma | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hypofractionated Radiotherapy for Soft Tissue Sarcoma (Experimental): Participants will be treated with 3-8 fractions, with the maximum prescribed dose to the Planning Tumor Volume (PTV) volume being 60 Gy delivered over a period of at most 8 weeks.
  Interventions: Radiation: Hypofractionated Radiotherapy

INTERVENTIONS:
Radiation: Hypofractionated Radiotherapy — Hypofractionated radiation is delivered using highly conformal technique, allowing for a high dose of radiation to be delivered precisely.

SUMMARY:
One of the main challenges in treating sarcomas with radiation is the toxicity to normal structures around the sarcoma. Early reports suggest Hypofractionated Radiotherapy will be safe and effective for treatment of soft tissue sarcomas. However, given the rarity of this disease, the diversity of histological sub-types, and the variety of locations where these can occur (anywhere in the body), more data is needed to provide understanding of the safety and efficacy of hypofractionated radiotherapy for treatment of this disease. The hypothesis is that by using hypofractionated radiotherapy, highly conformal high dose radiation can be delivered to soft tissue sarcomas, while respecting established normal tissue constraints and that local control rates will be greater than historical rates reported with conventional fractionation.

Eligible participants with biopsy proven soft tissue sarcoma will be on study for up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven soft tissue sarcoma, either localized and inoperable/unresectable or metastatic, that is deemed by the treating physician to be targetable with hypofractionated radiotherapy.
* Participant refuses surgery or is aware that surgery is not recommended for them
* Karnofsky performance status > 60
* Able to understand and sign an informed consent form

Exclusion Criteria:

* Pregnant
* Chemotherapy or systemic anti-cancer treatment within the preceding two weeks
* Unable to undergo imaging or positioning necessary for radiotherapy planning
* Prior radiation therapy in the field that, at the discretion of the treating physician, prevents safe delivery of hypofractionated radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants with 2-year Local Control | up to 2 years
  The primary endpoint is 2-year local control, defined as the proportion of participants whose best response as determined per RECIST criteria using imaging is Complete Response (CR), Partial Response (PR), or Stable Disease (SD) out of all participants who have received at least one fraction. Local control will be reported with an exact 95% confidence interval (CI).

SECONDARY OUTCOMES:
Proportion of Participants with 2-year Local Control: Primary Site vs Metastatic Site | up to 2 years
  2-year local control rates will be reported separately for primary sites vs. metastatic sites with exact 95% CI.
Proportion of Participants with 5-year Local Control: Primary Site vs Metastatic Site | up to 5 years
  5-year local control rates will be reported separately for primary sites vs. metastatic sites with exact 95% CI.
Complete Response Rate | up to 5 years
  The complete response (CR) rate will be reported with an exact 95% CI.
Progression Free Survival | up to 5 years
  Progression free survival (PFS) defined with follow-up radiological assessment with PFS calculated from the point of start of hypofractionated radiotherapy to the point of recurrence or death. Participants without documented progression who are alive at last follow-up will be censored at the date of the last radiologic assessment. PFS will be estimated using the Kaplan-Meier method.
Overall Survival | up to 5 years
  Overall survival (OS) defined from the point of start of hypofractionated radiotherapy to the time of death or last follow-up if alive. Participants who are alive at last follow-up will be censored. OS will be estimated using the Kaplan-Meier method.
Incidence of Acute Toxicity | up to 8 weeks
  Tabulated by type and grade.
Incidence of Long Term Toxicity | up to 5 years
  Tabulated by type and grade.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Morris, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/